CLINICAL TRIAL: NCT03167970
Title: Evaluation of Performance Characteristics of Capsule Endoscopy With PillCam UGI Capsule Compared to Standard Endoscopy for Screening of Barrett's Esophagus: A Prospective Tandem Study
Brief Title: Evaluation of Performance Characteristics of Capsule Endoscopy With PillCam UGI Capsule Compared to Standard Endoscopy
Status: Completed | Type: Observational
Sponsor: Midwest Biomedical Research Foundation (Other)
Collaborators: Medtronic Spine LLC (Industry)
Responsible Party: Sponsor
Organization: Midwest Veterans' Biomedical Research Foundation (Other)
Other Study IDs: PS0084
Record Dates: First submitted 2017-04-04; First posted 2017-05-30 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Barrett Esophagus
MeSH Terms: conditions — Barrett Esophagus | interventions — Complementary Therapies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Pill cam and EGD: Patients in this arm is requested to swallow the esophageal capsule and then undergo standard EGD.
  Interventions: Device: Pill cam; Other: EGD

INTERVENTIONS:
Device: Pill cam — Patient is asked to swallow the esophageal capsule.
Other: EGD — Patient will undergo standard EGD

SUMMARY:
This study is to examine the benefits of newly designed capsule with enhanced frame rate and wide angle compared to standard endoscopy, which may help enhance detecting esophageal diseases that otherwise may have been out of vision in the standard endoscopy, ultimately decreasing healthcare costs.

DETAILED DESCRIPTION:
This is a pilot, single center, prospective, tandem study. All veteran patients with Barrett's esophagus scheduled for an upper EGD at Veterans Affairs Medical Center (Kansas City, MO, USA) for check-up of BE will be asked to swallow the pillcam prior to an EGD. A member of the research team will approach a potential subject to discuss participation in the study, including background of the proposed study, inclusion and exclusion criteria, benefits and risks of the procedures and follow-up. If this is of interest to the subject, the informed consent form is discussed and presented. The subject must sign the consent form prior to enrollment. This form will have prior approval of the study site's Institutional Review Board (IRB). Failure to obtain informed consent renders the subject ineligible for the study

Eligible subjects at the participating institution who meet the inclusion criteria for this study will be offered the opportunity to participate in this clinical trial. To ensure that subjects are approached for potential study participation without bias, a Subject Screening Log will be maintained. This Log will track the basic demographic information of each subject approached for clinical trial inclusion and the resulting reason for exclusion from the clinical study if applicable.

The duration of the study is expected to be approximately 12 months. Enrollment of Study patients will cease when approximately 20 patients have been enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients age: ≥ 18 years
* Patients with BE length ≥ 1cm undergoing upper endoscopy
* Willingness to undergo both unsedated, capsule endoscopy and conventional EGD
* Ability to provide written, informed consent and understand the responsibilities of trial participation

Exclusion Criteria:

* Coagulopathy with INR > 1.5, thrombocytopenia with platelet counts < 50,000
* Pregnant or planning a pregnancy during the study period
* Dysphagia
* Known esophageal diverticulum or stricture
* Swallowing disorder
* Known luminal, gastrointestinal stricture
* History of esophageal, gastric surgery
* Esophageal or GI motility disorder
* Subject has a known history of unresolved drug or alcohol dependency that would limit ability to comprehend or follow instructions related to informed consent, post-treatment instructions, or follow-up guidelines
* Known or suspected gastrointestinal obstruction, strictures, or fistulas based on the clinical picture or pre-procedure testing and profile.
* Subjects with cardiac pacemakers or other implanted electromedical devices.
* Anticipated magnetic resonance imaging within 1 week of capsule ingestion

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a pilot, single center, prospective, tandem study. All veteran patients with Barrett's esophagus scheduled for an upper EGD at Veterans Affairs Medical Center (Kansas City, MO, USA) for check-up of BE will be asked to swallow the pillcam prior to an EGD.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2018-01-14 (Actual)

PRIMARY OUTCOMES:
The overall diagnostic accuracy of capsule endoscopy in predicting the presence and extent of Barrett's esophagus in comparison to standard esophagogastroduodenoscopy | 1 year
  The ability to accurately predict the presence of Barrett's esophagus by capsule endoscopy and standard EGD will be measured.

SECONDARY OUTCOMES:
Incidence of Treatment related adverse events of capsule endoscopy in comparison to standard esophagogastroduodenoscopy | 1 year
  Wireless capsule endoscopy is generally considered safe. Potential risks resulting from capsule endoscopy are reported low and may include discomfort while swallowing, accidental aspiration and capsule retention leading to small bowel obstruction and perforation. the investigator will measure tolerability of capsule endoscopy as well as standard endoscopy using visual analogue scale.

CONTACTS AND LOCATIONS:
Overall Officials: Prateek Sharma, MD, Principal Investigator — Kansas City VA Hospital
Locations (1):
- Kansas City VA Medical Center, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
This is a funded study. A copy of de-identified data set will be provided to the sponsor in the form of case report forms (CRF) at the end of the study.

REFERENCES:
- [Background] Sharma P. Clinical practice. Barrett's esophagus. N Engl J Med. 2009 Dec 24;361(26):2548-56. doi: 10.1056/NEJMcp0902173. No abstract available. PMID 20032324
- [Background] Eliakim R, Sharma VK, Yassin K, Adler SN, Jacob H, Cave DR, Sachdev R, Mitty RD, Hartmann D, Schilling D, Riemann JF, Bar-Meir S, Bardan E, Fennerty B, Eisen G, Faigel D, Lewis BS, Fleischer DE. A prospective study of the diagnostic accuracy of PillCam ESO esophageal capsule endoscopy versus conventional upper endoscopy in patients with chronic gastroesophageal reflux diseases. J Clin Gastroenterol. 2005 Aug;39(7):572-8. doi: 10.1097/01.mcg.0000170764.29202.24. PMID 16000923
- [Background] Chang JY, Talley NJ, Locke GR 3rd, Katzka DA, Schleck CD, Zinsmeister AR, Dunagan KT, Wu TT, Wang KK, Prasad GA. Population screening for barrett esophagus: a prospective randomized pilot study. Mayo Clin Proc. 2011 Dec;86(12):1174-80. doi: 10.4065/mcp.2011.0396. PMID 22134936